CLINICAL TRIAL: NCT03276260
Title: Evaluation of Medasense's PMD-200 During Surgery and Post Anesthesia Care
Status: Terminated | Type: Observational
Why Stopped: PI decided not to continue
Sponsor: Medasense Biometrics Ltd (Other)
Responsible Party: Sponsor
Other Study IDs: CLI-17-02
Record Dates: First submitted 2017-08-02; First posted 2017-09-08 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Surgery; Nociceptive Pain; Postoperative Pain
MeSH Terms: conditions — Nociceptive Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PMD-200 — Patient will be connected to PMD-200 by finger-probe before induction of anesthesia or sedation. Recording will continue during surgery until extubation or awakening. Recording will be initiated again as soon as the patient arrives to the PACU until discharge to the surgical ward or home.

SUMMARY:
Medasense's Pain Monitoring Device (PMD) is a novel non-invasive, bedside stand alone, continuous monitor that is designed to provide real-time information about changes in the nociception level of patients under general anesthesia during surgical procedures.

The PMD-200 System is based on real-time data acquisition and processing of physiological signals. The system displays the NOL index (a single numerical index) which is computed from recorded physiological parameters based on a proprietary algorithm.

DETAILED DESCRIPTION:
The aim of this observational study is to evaluate the pattern of the NOL index during surgery in the anesthetized patient and during the post-operative period in the awake patient.

Up to 100 patients scheduled for elective surgery under general, regional and local anesthesia and sedation, who meet all the inclusion and none of the exclusion criteria, will be enrolled after signing informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age 18 - 75 years
* ASA physical status 1-3
* Elective surgery

Exclusion Criteria:

* History of severe cardiac arrhythmia
* Abuse of alcohol or illicit drugs
* Preoperative opioid consumption for > 1 week
* History of mental retardation or any mental disease diagnosis
* Under sedation protocol - Patients with difficult spontaneous ventilation ( for e.g. patients with sleep apnea) will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 100 patients scheduled for elective surgery under general, regional and local anesthesia and sedation, who meet all the inclusion and none of the exclusion criteria, will be enrolled after signing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
The ability of NOL index to change in response to noxious and non noxious stimuli as well as in response to analgesic administration. | At time of surgery. 1 minute before and 1 minute after painful stimuli (for instance: intubation, skin incision, trocar insertion
Specificity and sensitivity of the NOL index for detecting nociception as evaluated by receiver operating characteristics curve (ROC) analysis. | At time of surgery, between the anaesthesia induction and extubation.
  The calculated area under the graph of change in NOL values in response to a painful stimulus, as mentioned in Outcome 1.

SECONDARY OUTCOMES:
The change in NOL Index in response to pre-defined non noxious and noxious stimuli during surgery in the anesthetized patient. | At time of surgery: pre-defined non noxious period - a period of 2 minutes with no noxious event with a minimal time period of 3 min prior and following laryngoscopy and intubation, skin incision or first trocar insertion.
  Pre-defined noxious events - laryngoscopy and intubation, skin incision or first trocar.
The change in NOL index in response to administration of analgesics. | At time of surgery, 1min before versus 1 min after administration of analgesics drugs.
Total fentanyl administration during surgery and anaesthesia and frequency of bolus administration. | At time of surgery, between the anaesthesia induction and extubation.
Total time with mean arterial pressure (MAP) < 65 mmHg and correlation to NOL values during surgery and anaesthesia. | At time of surgery, between the anaesthesia induction and extubation.
Total analgesics administration during PACU (arrival to discharge) and frequency of administration | Throughout PACU (Post Anesthesia Care Unit) stay, between entering PACU to discharge, an average of 2.5 hours.
NOL values during stay in PACU in the awake patient (arrival to discharge) | Throughout PACU (Post Anesthesia Care Unit) stay, between entering PACU to discharge, an average of 2.5 hours.
  The NOL will be calculated via the investigational device.
Patients' NRS (numerical rating scale ) values during stay in PACU (arrival to discharge). | Throughout PACU (Post Anesthesia Care Unit) stay, between entering PACU to discharge, an average of 2.5 hours.
  NRS will be recorded every 15 min in the PACU
Sedation scores during stay in PACU (arrival to discharge). | Throughout PACU (Post Anesthesia Care Unit) stay, between entering PACU to discharge, an average of 2.5 hours.
  Sedation scores will be recorded every 30 min in the PACU
Time to first analgesic request or administration in PACU. | Throughout PACU (Post Anesthesia Care Unit) stay, between entering PACU to discharge, an average of 2.5 hours.
Number of opioid adverse effects in PACU (nausea and vomiting, pruritus, desaturation, respiratory depression, apnea). | Throughout PACU (Post Anesthesia Care Unit) stay, between entering PACU to discharge, an average of 2.5 hours.
Time of readiness to discharge from PACU | Throughout PACU (Post Anesthesia Care Unit) stay, between entering PACU to discharge, an average of 2.5 hours.
  This time will be recorded since it may be different from the actual time of discharge which may be prolonged due to non-medical reasons.
The correlation between NOL values during surgery and anesthesia to NOL values during the post-operative period. | From the anaesthesia induction till the discharge from the PACU, an average of 5-6 hours.
  The NOL will be calculated via the investigational device.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Edry, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edry R, Recea V, Dikust Y, Sessler DI. Preliminary Intraoperative Validation of the Nociception Level Index: A Noninvasive Nociception Monitor. Anesthesiology. 2016 Jul;125(1):193-203. doi: 10.1097/ALN.0000000000001130. PMID 27171828
- [Background] Martini CH, Boon M, Broens SJ, Hekkelman EF, Oudhoff LA, Buddeke AW, Dahan A. Ability of the nociception level, a multiparameter composite of autonomic signals, to detect noxious stimuli during propofol-remifentanil anesthesia. Anesthesiology. 2015 Sep;123(3):524-34. doi: 10.1097/ALN.0000000000000757. PMID 26154185
- [Background] Treister R, Kliger M, Zuckerman G, Aryeh IG, Eisenberg E. Differentiating between heat pain intensities: the combined effect of multiple autonomic parameters. Pain. 2012 Sep;153(9):1807-1814. doi: 10.1016/j.pain.2012.04.008. Epub 2012 May 29. PMID 22647429
- [Background] Ben-Israel N, Kliger M, Zuckerman G, Katz Y, Edry R. Monitoring the nociception level: a multi-parameter approach. J Clin Monit Comput. 2013 Dec;27(6):659-68. doi: 10.1007/s10877-013-9487-9. Epub 2013 Jul 9. PMID 23835792